CLINICAL TRIAL: NCT05553197
Title: Intersession Processes in Psychotherapeutic Treatments Using an Ecological Momentary Assessment Approach (ISA-Bell)
Acronym: ISA-Bell
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Birgit Watzke (Other)
Collaborators: Universität Tübingen (Other)
Responsible Party: Sponsor-Investigator, Birgit Watzke, Full Professor, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10001C_200760
Record Dates: First submitted 2022-08-18; First posted 2022-09-23 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Depression
Keywords: Depression; Psychotherapy; Monitoring; Randomised Controlled Trial
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy; Ecological Momentary Assessment

STUDY DESIGN:
Intervention Model Description: 4/7 of participants will be randomised to CBT + EMA and 3/7 to TAU. This randomisation ratio is chosen to foster longitudinal analyses in the CBT + EMA group. Randomisation is stratified by pre-treatment severity of depressive symptoms. Participants with PHQ-9 scores 5-9 will be randomised separately from participants with PHQ-9 scores 10-20.
Masking Description: As is common in psychotherapy research, participants and care providers cannot be blinded to the intervention. Only subjective outcomes (i.e., participant-rated) are assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavior Therapy + Ecological Momentary Assessment (CBT + EMA) (Experimental): Cognitive Behavior Therapy + Ecological Momentary Assessment
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT); Other: Ecological Momentary Assessment (EMA)
- Treatment as Usual (TAU) (Active Comparator): Cognitive Behavioural Therapy (Treatment as Usual)
  Interventions: Behavioral: Cognitive Behavioural Therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy (CBT) — 20 sessions of face-to-face, individual CBT
Other: Ecological Momentary Assessment (EMA) — Two four-week blocks of twice daily ecological momentary assessment (EMA) of symptoms and inter-session processes
  Arms: Cognitive Behavior Therapy + Ecological Momentary Assessment (CBT + EMA)

SUMMARY:
The effects of a monitoring intervention as an add-on to face-to-face Cognitive Behavioral Therapy (CBT) for depression are assessed in this randomised trial. Monitoring consists of Ecological Momentary Assessment (EMA) of symptoms and inter-session processes via mobile phones. Twenty sessions of face-to-face CBT + EMA are compared to twenty sessions of face-to-face CBT (treatment as usual, TAU). 84 patients with mild to moderate depression will be randomised to CBT + EMA or to TAU.

DETAILED DESCRIPTION:
As mobile technologies advance, healthcare is increasingly utilising mobile interventions to accompany traditional interventions such as psychotherapy. Mobile assessments of symptoms and other processes are also used as low-level interventions and are believed to lead to symptom improvements in patients with symptoms of depression, for example. However, robust evidence on the health benefits of monitoring interventions in patients with depression is lacking.

The investigators are interested in the potential benefits of a monitoring intervention as an add-on to face-to-face Cognitive Behavioral Therapy (CBT) for depression. Therefore, the investigators will conduct a randomised trial to investigate the effects of a monitoring intervention consisting of Ecological Momentary Assessment (EMA) of symptoms and inter-session processes via mobile phones. Twenty sessions of face-to-face CBT + EMA will be compared to twenty sessions of face-to-face CBT (treatment as usual, TAU). Participants in the CBT + EMA group will be asked to answer monitoring questions twice daily for two four-week blocks during the CBT treatment. A total of 84 participants with mild to moderate depression will be randomized. Of these, 48 participants will be randomized to CBT + EMA and 36 participants will be randomized to TAU. The primary outcome of interest is change in the Patient Health Questionnaire (PHQ-9) score at four-month follow-up assessment.

Throughout the study, there will be five assessment timepoints: Baseline (before the first therapy session), four weeks after the fourth therapy session, four weeks after the twelfth therapy session, after the last session (post-treatment) and the 4-month follow-up (four months after the last therapy session).

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis of mild or moderate depression, first or recurrent episode (F32.0, F32.1, F33.0, F33.1)
* PHQ-9 ≥ 5
* Possession of smartphone with internet access
* Signed informed consent

Exclusion Criteria:

* Acute or past suicidality; self-reported
* Acute addiction (F10 - F19)
* Dysthymia (F34.1), postpartum depression, or severe depression (F32.3; F33.3)
* PHQ-9 > 20
* Depression not main mental health concern
* Planned onset or planned change in antidepressant medication
* History of psychotic symptoms, bipolar disorder, personality disorders, or organic brain disorders
* Cognitive impairment or physical disability that would hinder psychotherapy or the use of a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 4-month follow-up
  Participant-reported measure assessing depressive symptomatology. The total score of this nine-item scale ranges from 0-27, with higher scores indicating greater depression-symptom severity.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline, 4 weeks after the 4th session, 4 weeks after the 12th session, immediately after the last session and the 4-month follow-up
  Participant-reported measure assessing depressive symptomatology. The total score of this nine-item scale ranges from 0-27, with higher scores indicating greater depression-symptom severity.
Beck's Depression Inventory (BDI-II) | Baseline, 4 weeks after the 4th session, 4 weeks after the 12th session, immediately after the last session and the 4-month follow-up
  Participant-reported measure assessing changes in depressive symptoms. The total score of this twenty-one-item scale ranges from 0-63, with higher scores indicating greater depression severity.
Certainty About Mental States Questionnaire (CAMSQ) | Baseline, 4 weeks after the 4th session, 4 weeks after the 12th session, immediately after the last session and the 4-month follow-up
  Participant-reported measure assessing mentalisation of oneself and others. The total score of this forty-item scale ranges from 40-280, with higher scores indicating a greater frequency of successful mentalisation.
Dysfunctional Attitude Scale (DAS-18A) | Baseline, 4 weeks after the 4th session, 4 weeks after the 12th session, immediately after the last session and the 4-month follow-up
  Participant-reported measure assessing dysfunctional attitudes. The total score of this eighteen-item scale ranges from 18-126, with higher scores indicating greater levels of dysfunctional attitudes.
Depression-Specific Self-Efficacy Expectation Questionnaire (DSWE) | Baseline, 4 weeks after the 4th session, 4 weeks after the 12th session, immediately after the last session and the 4-month follow-up
  Participant-reported measure assessing depression-specific self-efficacy. The total score of this five-item scale ranges from 0-25, with higher scores indicating greater levels of depression-specific self-efficacy.
Evaluation of Treatment Progress Questionnaire (FEP-2) | Baseline, 4 weeks after the 4th session, 4 weeks after the 12th session, immediately after the last session and the 4-month follow-up
  Participant-reported measure assessing subjective treatment progress. The total score of this forty-item scale ranges from 40-200, with higher scores indicating poorer treatment outcome.
Level of Personality Functioning Scale - Brief Form (LPFS-BF 2.0) | Baseline, 4 weeks after the 4th session, 4 weeks after the 12th session, immediately after the last session and the 4-month follow-up
  Participant-reported measure assessing the level of personality functioning. The total score of this twelve-item scale ranges from 12-48, with higher scores indicating lower levels of functioning.
Positive and Negative Affect Schedule (PANAS) | Baseline, 4 weeks after the 4th session, 4 weeks after the 12th session, immediately after the last session and the 4-month follow-up
  Participant-reported measure assessing positive and negative affect using two subscales. The total score of each 10-item-subscale ranges from 10-50 with higher scores indicating greater levels of positive or negative affect in the corresponding subscales.
Personality Inventory for DSM-5 - Brief Form Plus (PID-5-BF+ M) | Baseline, 4 weeks after the 4th session, 4 weeks after the 12th session, immediately after the last session and the 4-month follow-up
  Participant-reported measure assessing personality traits. The total score of this thirty-six-item scale ranges from 0-108, with higher scores indicating greater personality pathology.
Health Survey - Short Form (SF-8) | Baseline, 4 weeks after the 4th session, 4 weeks after the 12th session, immediately after the last session and the 4-month follow-up
  Participant-reported measure assessing changes in health-related quality of life.The total score of this eight-item scale ranges from 8-42, with higher scores indicating poorer health-related quality of life.
Symptoms Checklist (SCL-K-9) | Baseline, 4 weeks after the 4th session, 4 weeks after the 12th session, immediately after the last session and the 4-month follow-up
  Participant-reported measure assessing symptoms during psychotherapy. The total score of this nine-item scale ranges from 0-36, with higher scores indicating greater symptom severity.
Treatment Satisfaction Questionnaire (ZUF-8) | Immediately after the last session
  Participant-reported measure assessing patients' satisfaction with treatment. The total score of this eight-item scale ranges from 8-32, with higher scores indicating greater treatment satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Watzke, PhD, Principal Investigator — University of Zurich
Locations (1):
- Psychotherapeutisches Zentrum Universität Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No